CLINICAL TRIAL: NCT07216261
Title: Implementing Cognitive Behavioral Therapy for Insomnia With Older Veterans: Function QUERI 3.0 (QUE 25-008)
Brief Title: Implementing Cognitive Behavioral Therapy for Insomnia (SWELL): Function QUERI 3.0
Acronym: SWELL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 25-004
Record Dates: First submitted 2025-10-02; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Insomnia
Keywords: Sleep Disorders; Implementation Science; Functional Status; Quality of Life; Cognitive Behavioral Therapy; Veterans
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized trial (parallel-CRT): used in pragmatic evaluations of health program or policy interventions, where half the clusters (in this case, VA sites) are randomly assigned to one of two interventions: Foundational support only (active comparator) vs. Foundational support plus Reach+Equity Implementation Bundle (experimental).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foundational Support (Active Comparator): Foundational Support uses the Replicating Effective Program (REP) implementation strategy and includes 5 elements that were developed and tested in our prior Function QUERI work: shareholder engagement, SWELL toolkit, online shared resources (SharePoint) access for clinical program training materials, data reports to assist sites with tracking their data, and Diffusion Networks to promote peer-to-peer sharing and implementation support.
  Interventions: Other: Implementation Strategy: Foundational Support
- Reach+Equity Bundle (Experimental): The Reach+Equity bundle will include the same activities as foundational support plus the Reach+Equity bundle activities which include: 1) external facilitation (designed to provide an outside perspective to help sites identify barriers, develop effective strategies, and navigate complex change processes particularly through the lens of achieving equitable reach); 2) equity in implementation toolkit (guide that supports awareness and consideration of equitable program reach and delivery during the implementation process); and 3) equity-focused data-driven monitoring (inform progress regarding equitable reach-related goals).
  Interventions: Other: Implementation Strategy: Reach+Equity Bundle

INTERVENTIONS:
Other: Implementation Strategy: Foundational Support — The primary goal of SWELL is to compare implementation approaches while also gathering information on clinical effectiveness of the EBP in its new context. All sites will be randomized to receive 1) foundational REP implementation support alone or 2) foundational REP and Reach+Equity. We propose that low intensity implementation support that promotes engagement with SWELL (defined as foundational support), will be sufficient for some but not all facilities to successfully incorporate SWELL into routine practice.
  Other Names: Foundational REP
  Arms: Foundational Support
Other: Implementation Strategy: Reach+Equity Bundle — We hypothesize that adding the Reach+Equity bundle to foundational REP, compared to foundational REP alone, will result in superior implementation outcomes.
  Other Names: Enhanced Support
  Arms: Reach+Equity Bundle

SUMMARY:
Implementing Cognitive Behavioral Therapy for Insomnia with Older Veterans (SWELL): Function QUERI 3.0 aims to compare implementation approaches while also gathering information on clinical effectiveness of the EBP in its new context. The overall goal is to address a key priority within the implementation science field - identifying and refining metrics for equity and impact. The overall goal is to implement, evaluate, and sustain SWELL in 20 VA facilities using a type III effectiveness-implementation hybrid study framework and parallel CRT design.

DETAILED DESCRIPTION:
Background/Purpose. As many as two-thirds of older Veterans meet criteria for chronic insomnia disorder, defined as three or more months of subjective complaints related to difficulty falling or staying asleep or waking too early and/or poor nighttime sleep associated with daytime impairment. Left untreated, chronic insomnia can negatively impact quality-of-life and contribute to accelerated cognitive and functional decline.

CBTI is the recommended first-line treatment for chronic insomnia; however, despite several VA initiatives focused on the scale-up of CBTI, fewer than 5% of older Veterans with chronic insomnia have received this evidence-based therapy. To address this challenge, the team adapted CBTI for older Veterans. In a series of trials to evaluate the adapted program, Sleep Well, Live Well (SWELL), the team found significant improvements in nighttime sleep and daytime functioning that lasted up to one year after the end of treatment. Notably, using a comprehensive training and supervision model, these studies demonstrated that non-psychologists can effectively deliver CBTI. The investigators' evidence-based and age-friendly CBTI program, SWELL, involves five sessions delivered weekly with a trained provider. Content focuses on establishing a regular sleep-wake schedule, moving non-sleep activities out of the bedroom, establishing healthy sleep habits, relaxation near bedtime, and addressing unhealthy expectations about sleep.

Objectives. The investigators plan to develop scalable approaches to implement and sustain SWELL as well as evaluate reach with foundational support versus the enhanced implementation strategy (Reach+Equity bundle).

Key questions. How can the Reach+Equity bundle be optimized? What are shareholder perspectives on the refinements needs for SWELL foundational activities, as well as strategies to enhance equitable reach (Reach+Equity bundle)? Are there differences in implementation outcomes (reach, fidelity, adoption, cost) at six, 12, and 18 months between arms? Is reach representative of Veterans experiencing chronic insomnia at participating sites (equitable reach) and does this differ between arms? Are there differences in effectiveness outcomes (insomnia severity, function) between arms? How do sites experience implementation strategies in each arm? To address the question: Are there differences in implementation outcomes (reach [primary], fidelity, adoption) between arms? The investigators will use generalized linear models to examine the effect of foundational REP vs. Reach+Equity on implementation outcomes of reach and fidelity at 6, 12, and 18-months (primary). The investigators will examine how implementation outcomes change over time using descriptive methods (e.g. plots, descriptive statistics, subgroups). The investigators will compare average time to adoption between study arms. The investigators will examine equitable reach by calculating participation to prevalence ratios (PPRs) by site and implementation arm. The investigators will explore ratios by rurality and gender as well as race, sex and age. To address the question: Are there differences in effectiveness outcomes (insomnia symptoms, function) between arms, the investigators will describe effectiveness outcomes for patients who initiate the SWELL program, overall and by study arm. The investigators will calculate change in patient outcomes based on patients' pre- and post-program visits. Generalized linear mixed effect models including all time points for patient outcomes will be fit to account for clustering of patients within site and repeated measures of patient outcomes.

Methodology. To evaluate implementation, the investigators will randomize sites (n=20) 1:1 to either foundational support or foundational support plus the Reach+Equity bundle. The investigators will use generalized linear models to examine the effect of foundational vs. Reach+Equity on implementation outcomes at 18-months.

ELIGIBILITY:
Inclusion Criteria:

* meet diagnostic criteria for chronic insomnia disorder (with or without documented diagnosis)
* absence of a CBTI contraindication

  * i.e., comorbid condition that makes CBTI unsafe), including uncontrolled seizure disorders, bipolar disorder I, and/or too medically or psychiatrically unstable to engage in a multi-session treatment
  * patients can be referred to SWELL by a clinician or self-referred

Exclusion Criteria:

* younger than 60
* do not meet criteria for enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach | 18 months
  Reach (primary) will be defined as the number of older Veterans who initiate SWELL at six, 12, and 18 (primary) months.

SECONDARY OUTCOMES:
Fidelity | 18 months
  Fidelity will be defined as the mean number of SWELL sessions completed per enrolled older Veteran.
Adoption | 18 months
  Adoption will be defined as delivering the program to ≥5 unique Veterans.

OTHER OUTCOMES:
Cost of Treatment | 18 months
  Budget impacts will be assessed using implementation process data (e.g. office hours, Diffusion Network, and facilitation call notes) and VA salary and managerial cost accounting data to describe EBP delivery costs and to calculate the costs of the two implementation approaches (foundational REP and Reach+Equity). Two types of costs will be collected for each site using brief monthly surveys to track implementation activities: (1) clinical delivery team costs incurred; and (2) implementation strategy costs incurred. Unlike in a cost-effectiveness analysis evaluating two distinct treatments, the investigators will not evaluate healthcare costs because all individual participants will receive the same clinical treatment regardless of a site's implementation strategy.
Insomnia Severity | Baseline
  Mean score on Insomnia Severity Index (ISI). This 7-item scale measures self-reported severity of insomnia symptoms.
  Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
Insomnia Severity | 6 weeks
  Mean score on Insomnia Severity Index (ISI). This 7-item scale measures self-reported severity of insomnia symptoms.
  Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Hughes, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Jennifer L Martin, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format. Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication. No data or statistical code that could lead to re-identification of individuals will be released. Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form. The statistician will create de-identified, publication-specific datasets that includes variables from statistical models presented in publication. Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.
Supporting Information: Study Protocol
Time Frame: Available upon request.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.
URL: https://www.durham.hsrd.research.va.gov/Function_Independence_QUERI.asp